CLINICAL TRIAL: NCT05757908
Title: An Open-Label, Single-Arm Study in Moderate Asthma Participants Comparing the Treatment With Long-Acting Beta Agonist Between At-Home Mobile Spirometry and In-Clinic Spirometry (LEARN)
Brief Title: Study Comparing At-Home Mobile Spirometry to In-Clinic in Moderate Asthma Participants Taking Long-Acting Beta Agonist
Acronym: LEARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koneksa Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KH008
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Moderate Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Long-Acting Beta Agonist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long-Acting Beta Agonist (Other): Standard of care LABA
  Interventions: Drug: Long-Acting Beta Agonist

INTERVENTIONS:
Drug: Long-Acting Beta Agonist — The Investigator will prescribe standard of care LABA to eligible study participants. Participants will self-administer LABA once or twice daily at the maximum feasible standard of care dosage, per the time points specified in the study Schedule of Assessments. LABA should be taken within 1 to 3 hours prior to morning and evening at-home mobile Spirometry testing.
  Other Names: LABA

SUMMARY:
The goal of this interventional study is to compare at-home mobile spirometry to in-clinic spirometry in participants with moderate asthma while taking a long-acting beta agonist (LABA).

The main questions it aims to answer are:

* Do at-home mobile spirometry and in-clinic spirometry assessments show a similar treatment effect (measured changes in FEV1) with the addition of LABA?
* Is at-home mobile spirometry as accurate as in-clinic spirometry in showing treatment effects (changes in FEV1)?

Participants will be asked to:

* Take standard of care LABA treatment once or twice a day
* Complete at-home mobile spirometry testing twice a day
* Complete asthma questionnaires twice a day
* Complete device use questionnaires
* Wear a wrist device (like a watch) to track physical activity and vital signs
* Visit the clinic for in-clinic spirometry testing once a week for 8 weeks

DETAILED DESCRIPTION:
The study will recruit up to 60 participants with moderate uncontrolled asthma who are taking inhaled corticosteroids (ICS) at the time of study enrollment but will require LABA treatment as judged by their treating physician. The study will assess the LABA treatment effect in clinic and mobile spirometry, assess the relationship between different readouts of mobile spirometry in addition to assessing asthma control as measured by ACQ-6, patient reported outcome questionnaire. Additional objectives include an evaluation of patient and site-specific satisfaction with mobile spirometry technology.

The study consists of a one-week screening period, one-week baseline period, and up to 6-week interventional assessment period consisting of addition of LABA, for an estimated participant duration of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 18 years or older
2. Body mass index (BMI) 18 - 40 mg/m2 inclusive
3. Participant with a diagnosis of moderate uncontrolled asthma
4. Participant must be using a medium to high daily dose of inhaled corticosteroids (ICS) for a minimum of 6 weeks prior to screening
5. Asthma that is not currently using long-acting beta-agonists (LABA) or log-acting muscarinic antagonist (LAMA) (ACQ score of 0.75 or higher) Note: A 2-week LABA/LAMA washout period is allowed prior to screening
6. Pre-bronchodilator FEV1 ≥ 60% and ≤100% of the predicted normal values at screening
7. A documented positive response to the reversibility test at screening, defined as improvement in FEV1 ≥ 12% and ≥ 200 mL over baseline after a Short Acting Beta Agonist (SABA) standard of care dose. Documented historical reversibility of up to 6 weeks is allowed.
8. Participant is judged to be in good health based on medical history, physical examination, and vital sign measurements
9. Non-smokers or ex-smokers (including vape or inhaled cannabis) who have stopped smoking more than 1 year ago
10. Women of childbearing potential must have a negative urine pregnancy test before enrolling at Baseline Day 1
11. Participant demonstrated ability to perform satisfactory in-clinic and at-home Spirometry according to ATS/ERS standards, as well as the mobile application to synchronize Spirometry data collection and respond to questionnaires during the Screening coaching/training period

Exclusion Criteria:

1. History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest and/or hypoxic seizures or hospitalization (including ER visits) for the treatment of asthma within 3 months prior to screening, or have been hospitalized or have attended the ER for asthma more than twice in prior 6 months
2. Occurrence of asthma exacerbations or respiratory tract infections within 4 weeks prior to Screening
3. History of substance abuse in the last 6 months, excluding medical or recreational non- inhaled marijuana
4. Currently taking other biologics to control asthma symptoms (allergy shots are acceptable)
5. Diagnosis of any other airway/pulmonary disease such as Chronic Obstructive Pulmonary Disease (COPD) as defined by the current Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines; or other lung diseases (e.g., emphysema, idiopathic pulmonary fibrosis, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency or restrictive lung disease)
6. Clinically unstable participants or history of non-compliance as assessed by the PI
7. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 1 month prior to screening
8. Participant has a history of neoplastic disease. Exceptions: Participants with (1) an adequately treated basal or squamous cell carcinoma or carcinoma in situ of the cervix; (2) localized or regional prostate cancer; other malignancies which have been successfully treated > 5 years prior to screening without evidence of recurrence may participate
9. Participants treated with oral or parenteral corticosteroids in the previous 4 weeks prior to screening
10. You may not be able to participate in this study if you have been in another investigational drug study for 30 days prior to this study unless approval is given from the Sponsor. Additionally, you cannot be involved in another investigational drug study during your participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Measured FEV1 Change to Treatment Effect | Baseline Day 1 through Day 43 End of Study
  Detection of treatment effect as measured by change from baseline in morning FEV1 measured in change over time for at-home mobile and in-clinic Spirometry
Measured FEV1 Change and Comparison of Variability | Baseline Day 1 through Day 43 End of Study
  Change from baseline and comparison of variability (measured via confidence interval) in morning FEV1 for at-home morning mSpirometry compared to morning in-clinic Spirometry

SECONDARY OUTCOMES:
Mobile Spirometry Compliance | Baseline Day 1 through Day 43 End of Study
  Percentage of compliance for once and twice daily at-home mSpirometry
Relationship Between In-clinic and Mobile Spirometry Parameters | Baseline Day 1 through Day 43 End of Study
  1. Evaluate the relationship between in-clinic and mSpirometry FEV1 and other Spirometry parameters (e.g., FVC)
  2. Relationship between other Spirometry measurements (e.g., FVC)
Diurnal Differences in Mobile Spirometry | Baseline Day 1 through Day 43 End of Study
  Diurnal differences in morning versus evening for at-home mSpirometry parameters, e.g., FEV1
Time to Treatment Effect | Baseline Day 1 through Day 43 End of Study
  Time to treatment effect detection using at-home mSpirometry via change in FEV1
Treatment Effect | Baseline Day 1 through Day 43 End of Study
  Treatment effect as measured by change from baseline in ACQ-6
Mobile Spirometry Changes | Baseline Day 1 through Day 43 End of Study
  Relationship between at-home mSpirometry changes and changes in ACQ-6
Device Use Surveys | Baseline Day 1 through Day 43 End of Study
  1. Site clinical care team likelihood to recommend at-home mSpirometry
  2. Site clinical care team ease-of-use of at-home mSpirometry
  3. Site clinical care team device satisfaction
  4. Participant likelihood to recommend at-home mSpirometry
  5. Participant ease-of-use of at-home mSpirometry
  6. Participant device satisfaction

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - AllerVie Research Clinic, Birmingham, Alabama
  - AllerVie Research Clinic, Columbus, Georgia
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - The Asthma & Allergy Center, PC, Bellevue, Nebraska
  - American Health Research, Charlotte, North Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - El Paso Pulmonary Association, El Paso, Texas
  - South Texas Allergy & Asthma Medical Professionals Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Izmailova ES, Kilian R, Bakker JP, Evans S, Scotina AD, Reiss TF, Singh D, Wagner JA. Study protocol: A comparison of mobile and clinic-based spirometry for capturing the treatment effect in moderate asthma. Clin Transl Sci. 2023 Nov;16(11):2112-2122. doi: 10.1111/cts.13615. Epub 2023 Sep 8. PMID 37602889